CLINICAL TRIAL: NCT00789672
Title: A Pilot Study to Evaluate Levodopa as Treatment for Residual Amblyopia in 8 to 17 Year Olds
Brief Title: Pilot Study to Evaluate Levodopa as Treatment for Residual Amblyopia
Acronym: ATS14
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Jaeb Center for Health Research (Other)
Collaborators: National Eye Institute (NEI) (NIH)
Responsible Party: Principal Investigator, Ray Kraker, Director, PEDIG Coordinating Center, Jaeb Center for Health Research
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: NEI-141; 2U10EY011751 (NIH)
Record Dates: First submitted 2008-10-27; First posted 2008-11-13 (Estimated); Results first posted 2011-03-23 (Estimated); Last update posted 2016-07-13 (Estimated); Status verified 2016-07

CONDITIONS: Amblyopia
Keywords: Amblyopia; Patching; Levodopa
MeSH Terms: conditions — Amblyopia | interventions — carbidopa, levodopa drug combination

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Lower Dose (3-1) levodopa/carbidopa (Active Comparator): Oral levodopa 0.51 mg/kg tid with carbidopa 0.17 mg/kg tid (3 to 1 formulation) combined with 2 hours of daily patching, with a rapid taper of medication before a primary outcome exam 9 weeks after starting medication.
  Interventions: Device: patching; Drug: levodopa/carbidopa
- Higher Dose (4.5-1) levodopa/carbidopa (Active Comparator): Oral levodopa 0.76 mg/kg tid with carbidopa 0.17 mg/kg tid (approximately 4.5 to 1 formulation) combined with 2 hours of daily patching, with a rapid taper of medication before a primary outcome exam 9 weeks after starting medication.
  Interventions: Drug: levodopa/carbidopa; Device: patching

INTERVENTIONS:
Drug: levodopa/carbidopa — Oral levodopa 0.76 mg/kg tid with carbidopa 0.17 mg/kg tid (approximately 4.5 to 1 formulation)
  Arms: Higher Dose (4.5-1) levodopa/carbidopa
Device: patching — 2 hours daily patching
  Other Names: Coverlet, 3M Opticlude, Ortopad®
Drug: levodopa/carbidopa — Oral levodopa 0.51mg/kg tid with carbidopa 0.17 mg/kg tid (3 to 1 formulation)
  Arms: Lower Dose (3-1) levodopa/carbidopa

SUMMARY:
This pilot study is being conducted as a prelude to a randomized trial to compare levodopa/carbidopa plus patching versus patching alone. The purpose of the pilot study is to demonstrate recruitment potential, to provide prospective data on the tolerability of levodopa as a treatment for amblyopia, to provide limited data on its safety, to provide limited data on it's efficiency, and to provide data to assist in selecting a dose to use in a subsequent phase 3 randomized trial. In addition, this study will provide the opportunity for investigators to gain experience in using levodopa prior to a randomized trial.

DETAILED DESCRIPTION:
Amblyopia is the most common cause of monocular visual impairment in both children and young and middle-aged adults. Both patching and atropine are accepted treatment modalities for the management of moderate amblyopia in children. Despite best efforts with conventional amblyopia treatment, many older children and teenagers with amblyopia fail to achieve normal visual acuity in the amblyopic eye. In a previous PEDIG study (ATS3) where children 7 to 13 years old were treated with atropine and patching, only 36% of the children with moderate amblyopia and only 23% of the children with severe amblyopia achieved 20/40 or better acuity.

ELIGIBILITY:
Inclusion Criteria:

* Age 8 to < 18 years old
* Amblyopia associated with strabismus, anisometropia, or both
* Visual acuity in the amblyopic eye 18 to 67 letters inclusive (20/50 to 20/400)
* Visual acuity in the sound eye ≥ 78 letters (20/25 or better)
* Current amblyopia treatment of at least 2 hours patching per day
* No improvement in best-corrected amblyopic eye visual acuity between two consecutive visits at least 4 weeks apart using the same testing method and optimal spectacle correction (if needed), with no improvement of more than 4 letters or one logMAR line.

Exclusion Criteria:

* Myopia more than -6.00 D (spherical equivalent) in either eye.
* Current vision therapy or orthoptics
* Ocular cause for reduced visual acuity

  • nystagmus per se does not exclude the subject if the above visual acuity criteria are met
* Prior intraocular or refractive surgery
* History of narrow-angle glaucoma
* Strabismus surgery planned within 16 weeks
* Known allergy to levodopa-carbidopa
* History of dystonic reactions
* Current requirement to take oral iron supplements including multivitamins containing iron during the 8 weeks of treatment with levodopa-carbidopa
* Current use of antihypertensive, anti-depressant medications, phenothiazines, butyrophenones, risperidone and isoniazid, non-specific monoamine oxidase inhibitors
* Current use of medication for the treatment of attention deficit hyperactivity disorder
* Known gastrointestinal or liver disease
* History of melanoma
* Known psychological problems
* Known skin reactions to patch or bandage adhesives
* Prior levodopa treatment
* Current treatment with topical atropine
* Females who are pregnant, lactating, or intending to become pregnant within the next 16 weeks.

  * A negative urine pregnancy test will be required for all females who have experienced menarche.
  * Requirements regarding the establishment of pregnancy and monitoring of pregnancy over the course of the study as defined by each individual Institutional Review Board may supersede these criteria.

Ages: 8 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 33 (Actual)
Dates: Start 2009-01; Primary Completion 2009-09 (Actual); Study Completion 2009-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael X. Repka, M.D., Study Chair — Wilmer Eye Institute
Locations (1):
- Wilmer Eye Institute, Baltimore, Maryland, United States

REFERENCES:
- [Result] Repka MX, Kraker RT, Beck RW, Atkinson CS, Bacal DA, Bremer DL, Davis PL, Gearinger MD, Glaser SR, Hoover DL, Laby DM, Morrison DG, Rogers DL, Sala NA, Suh DW, Wheeler MB; Pediatric Eye Disease Investigator Group. Pilot study of levodopa dose as treatment for residual amblyopia in children aged 8 years to younger than 18 years. Arch Ophthalmol. 2010 Sep;128(9):1215-7. doi: 10.1001/archophthalmol.2010.178. No abstract available. PMID 20837811

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Eligibility criteria included age 8 to <18 years, best-corrected visual acuity in the amblyopic eye between 67 and 18 letters inclusive measured with E-ETDRS, fellow eye best-corrected visual acuity of 78 letters or better, and the presence or history of strabismus and/or anisometropia.
Pre-assignment Details: At enrollment, subjects were required to have been treated with at least 2 hours of patching per day of daily patching and while on that therapy, have had stable visual acuity (5 letters or one logMAR line of improvement since a previous visit at least 8 weeks earlier)
Groups:
- Lower Dose 0.51 mg Levodopa/Carbidopa: Oral levodopa 0.51 mg/kg tid with carbidopa 0.17 mg/kg tid combined with 2 hours of daily patching, with a rapid taper of medication before a primary outcome exam.
- Higher Dose 0.76 mg Levodopa/Carbidopa: Oral levodopa 0.76 mg/kg tid with carbidopa 0.17 mg/kg tid combined with 2 hours of daily patching, with a rapid taper of medication before a primary outcome exam.
Period: Overall Study
Arm/Group | Lower Dose 0.51 mg Levodopa/Carbidopa | Higher Dose 0.76 mg Levodopa/Carbidopa
Started | 16 | 17
Completed | 16 | 17
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Lower Dose 0.51 mg Levodopa/Carbidopa | Higher Dose 0.76 mg Levodopa/Carbidopa | Total
Number analyzed (Participants) | 16 | 17 | 33
Age, Continuous [Mean (Standard Deviation); unit: years] | 11.3 (2.2) | 11.0 (2.2) | 11.1 (2.2)
Age, Customized [Number; unit: participants] — Age at enrollment in years
  participants
    8 to <9 | 3 | 3 | 6
    9 to <10 | 2 | 3 | 5
    10 to <11 | 3 | 4 | 7
    11 to <12 | 3 | 1 | 4
    12 to <13 | 0 | 3 | 3
    13 to <14 | 3 | 1 | 4
    14 to <15 | 2 | 0 | 2
    15 to <16 | 0 | 2 | 2
    16 to <17 | 0 | 0 | 0
    17 to <18 | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 | 9 | 19
  Male | 6 | 8 | 14
Region of Enrollment [Number; unit: participants]
  United States | 16 | 17 | 33
Cause of Amblyopia [Number; unit: participants]
  Strabismus | 2 | 5 | 7
  Anisometropia | 6 | 5 | 11
  Strabismus and anisometropia | 8 | 7 | 15
Distance Visual Acuity in Amblyopic Eye [Number; unit: participants] — Visual acuity was measured with the electronic early treatment diabetic retinopathy study (E-ETDRS) method and resulted in a letter score that could range from 0 to 97 letters, with 0 being the worst and 97 being the best. Letter scores are presented as Snellen Equivalents for presentation (i.e. 20/20 includes those with letter scores between 83 and 87 letters, 20/25 includes those with letter scores between 78 to 82 letters, etc.).
  participants
    20/400 (18 to 22 letters) | 0 | 1 | 1
    20/320 (23 to 27 letters) | 0 | 0 | 0
    20/250 (28 to 32 letters) | 0 | 1 | 1
    20/200 (33 to 37 letters) | 1 | 1 | 2
    20/160 (38 to 42 letters) | 1 | 1 | 2
    20/125 (43 to 47 letters) | 0 | 1 | 1
    20/100 (48 to 52 letters) | 2 | 0 | 2
    20/80 (53 to 57 letters) | 4 | 6 | 10
    20/63 (58 to 62 letters) | 4 | 5 | 9
    20/50 (63 to 67 letters) | 4 | 1 | 5
Distance Visual Acuity in Fellow Eye [Number; unit: participants] — Visual acuity was measured with the electronic early treatment diabetic retinopathy study (E-ETDRS) method and resulted in a letter score that could range from 0 to 97 letters, with 0 being the worst and 97 being the best. Letter scores are presented as Snellen Equivalents for presentation (i.e. 20/20 includes those with letter scores between 83 and 87 letters, 20/25 includes those with letter scores between 78 to 82 letters, etc.).
  participants
    20/25 (78 to 82 letters) | 4 | 4 | 8
    20/20 (83 to 87 letters) | 6 | 8 | 14
    20/16 (88 to 92 letters) | 5 | 5 | 10
    20/12 (93 to 97 letters) | 1 | 0 | 1
Race/Ethnicity [Number; unit: participants]
  White | 14 | 17 | 31
  African-American | 1 | 0 | 1
  Hispanic or Latino | 1 | 0 | 1
  Asian | 0 | 0 | 0
  More than one race | 0 | 0 | 0
  Unknown/Not reported | 0 | 0 | 0
Refractive Error in Amblyopic Eye (spherical equivalent/diopters) [Number; unit: participants] — Spherical equivalent in diopters defined from cycloplegic refraction as sphere plus half the cylinder value
  participants
    <0.00D | 0 | 1 | 1
    0 to < +1.00D | 1 | 2 | 3
    +1.00 to <+2.00D | 1 | 1 | 2
    +2.00 to <+3.00D | 2 | 2 | 4
    +3.00 to <+4.00D | 3 | 2 | 5
    greater than or equal to +4.00D | 9 | 9 | 18
Refractive Error in Fellow Eye (spherical equivalent/diopters) [Number; unit: participants] — Spherical equivalent in diopters defined from cycloplegic refraction as sphere plus half the cylinder value
  participants
    <0.00D | 1 | 0 | 1
    0 to < +1.00D | 6 | 10 | 16
    +1.00 to <+2.00D | 5 | 3 | 8
    +2.00 to <+3.00D | 2 | 3 | 5
    +3.00 to <+4.00D | 2 | 1 | 3
    greater than or equal to +4.00D | 0 | 0 | 0
Mean (SD) Distance Visual Acuity in Amblyopic Eye [Mean (Standard Deviation); unit: letters] — Visual acuity was measured with the electronic early treatment diabetic retinopathy study (E-ETDRS) method and resulted in a letter score that could range from 0 to 97 letters, with 0 being the worst and 97 being the best.
  letters | 56.2 (8.8) | 50.5 (12.2) | 53.2 (10.9)
Mean (SD) Distance Visual Acuity in Fellow Eye [Mean (Standard Deviation); unit: letters] — Visual acuity was measured with the electronic early treatment diabetic retinopathy study (E-ETDRS) method and resulted in a letter score that could range from 0 to 97 letters, with 0 being the worst and 97 being the best.
  letters | 86.4 (4.5) | 85.5 (3.3) | 85.9 (3.9)
Mean (SD) Intereye Acuity Difference [Mean (Standard Deviation); unit: letters] — Visual acuity was measured with the electronic early treatment diabetic retinopathy study (E-ETDRS) method and resulted in a letter score in each eye that could range from 0 to 97 letters. Intereye difference calculated as the difference in letters between the sound eye and amblyopic eye (positive difference indicates sound eye better).
  letters | 30.2 (11.7) | 35.1 (13.6) | 32.7 (12.7)
Mean (SD) Spherical Equivalent Refractive Error in Amblyopic Eye [Mean (Standard Deviation); unit: diopters] — Spherical equivalent in diopters defined from cycloplegic refraction as sphere plus half the cylinder value
  diopters | 4.05 (1.92) | 3.28 (1.93) | 3.65 (1.93)
Mean (SD) Spherical Equivalent Refractive Error in Fellow Eye [Mean (Standard Deviation); unit: diopters] — Spherical equivalent in diopters defined from cycloplegic refraction as sphere plus half the cylinder value
  diopters | 1.20 (1.17) | 1.04 (0.99) | 1.12 (1.07)
Weight in Kilograms [Median (Full Range); unit: kilograms] | 47 [25 to 71] | 34 [23 to 74] | 42 [23 to 74]

OUTCOME MEASURES:

1. Primary Outcome: Distribution of Amblyopic Eye Visual Acuity Letter Scores at 9 Weeks After Starting Levodopa
Description: Visual acuity was measured with the electronic early treatment diabetic retinopathy study (E-ETDRS) method and resulted in a letter score that could range from 0 to 97 letters, with 0 being the worst and 97 being the best. Letter scores are presented as Snellen Equivalents for presentation (i.e. 20/20 includes those with letter scores between 83 and 87 letters, 20/25 includes those with letter scores between 78 to 82 letters, etc.).
Time Frame: 9 weeks after starting levodopa
Measure: Number; unit: participants
Arm/Group | Lower Dose 0.51 mg Levodopa/Carbidopa | Higher Dose 0.76 mg Levodopa/Carbidopa
Number analyzed (Participants) | 16 | 17
participants
  <20/100 (<47 letters) | 2 | 5
  20/100 (47 to 52 letters) | 2 | 0
  20/80 (53 to 57) | 1 | 1
  20/63 (58 to 62) | 3 | 5
  20/50 (63 to 67) | 4 | 3
  20/40 (68-72 letters) | 3 | 2
  20/32 (73 to 77 letters) | 1 | 1

2. Primary Outcome: Mean Amblyopic Eye Visual Acuity Letter Scores at 9 Weeks After Starting Levodopa
Description: Visual acuity was measured with the electronic early treatment diabetic retinopathy study (E-ETDRS) method and resulted in a letter score that could range from 0 to 97 letters, with 0 being the worst and 97 being the best.
Time Frame: 9 weeks after starting levodopa
Measure: Mean (Standard Deviation); unit: letters
Arm/Group | Lower Dose 0.51 mg Levodopa/Carbidopa | Higher Dose 0.76 mg Levodopa/Carbidopa
Number analyzed (Participants) | 16 | 17
letters | 59.9 (9.7) | 56.5 (12.7)

3. Primary Outcome: Distribution of Change in Amblyopic Eye Visual Acuity Scores at 9 Weeks After Starting Levodopa
Description: Visual acuity was measured with the electronic early treatment diabetic retinopathy study (E-ETDRS) method and resulted in a letter score that could range from 0 to 97 letters, with 0 being the worst and 97 the best. A difference was calculated as the difference in letters between baseline and outcome with positive difference indicating improvement in acuity.
Time Frame: baseline to 9 weeks
Measure: Number; unit: participants
Arm/Group | Lower Dose 0.51 mg Levodopa/Carbidopa | Higher Dose 0.76 mg Levodopa/Carbidopa
Number analyzed (Participants) | 16 | 17
participants
  >=15 letters worse | 0 | 0
  10 to 14 letters worse | 0 | 0
  5 to 9 letters worse | 0 | 1
  Within plus or minus 4 letters | 9 | 5
  5 to 9 letters better | 5 | 6
  10 to 14 letters better | 2 | 4
  >=15 letters better | 0 | 1

4. Secondary Outcome: Distribution of Amblyopic Eye Visual Acuity Letter Scores at 4 Weeks After Enrollment
Description: Visual acuity was measured with the electronic early treatment diabetic retinopathy study (E-ETDRS) method and resulted in a letter score that could range from 0 to 97 letters, with 0 being the worst and 97 the best. Letter scores are presented as Snellen Equivalents for presentation (i.e. 20/20 includes those with letter scores between 83 and 87 letters, 20/25 includes those with letter scores between 78 to 82 letters, etc.).
Time Frame: 4 weeks after enrollment
Measure: Number; unit: participants
Arm/Group | Lower Dose 0.51 mg Levodopa/Carbidopa | Higher Dose 0.76 mg Levodopa/Carbidopa
Number analyzed (Participants) | 16 | 17
participants
  <20/100 (<47 letters) | 2 | 4
  20/100 (47 to 52 letters) | 2 | 1
  20/80 (53 to 57) | 1 | 3
  20/63 (58 to 62) | 4 | 5
  20/50 (63 to 67) | 4 | 3
  20/40 (68-72 letters) | 3 | 1
  20/32 (73 to 77 letters) | 0 | 0

5. Secondary Outcome: Mean Amblyopic Eye Visual Acuity Letter Scores at 4 Weeks Post Enrollment
Description: Visual acuity was measured with the electronic early treatment diabetic retinopathy study (E-ETDRS) method and resulted in a letter score that could range from 0 to 97 letters, with 0 being the worst and 97 the best.
Time Frame: 4 weeks after enrollment
Measure: Mean (Standard Deviation); unit: letters
Arm/Group | Lower Dose 0.51 mg Levodopa/Carbidopa | Higher Dose 0.76 mg Levodopa/Carbidopa
Number analyzed (Participants) | 16 | 17
letters | 59.1 (9.2) | 54.3 (12.9)

6. Secondary Outcome: Distribution of Amblyopic Eye Visual Acuity Letter Scores at 10 Weeks After Stopping Levodopa
Description: as for outcome 4
Time Frame: 10 weeks after stopping levodopa
Measure: Number; unit: participants
Arm/Group | Lower Dose 0.51 mg Levodopa/Carbidopa | Higher Dose 0.76 mg Levodopa/Carbidopa
Number analyzed (Participants) | 16 | 17
participants
  <20/100 (<47 letters) | 2 | 5
  20/100 (47 to 52 letters) | 0 | 1
  20/80 (53 to 57) | 3 | 2
  20/63 (58 to 62) | 4 | 3
  20/50 (63 to 67) | 2 | 6
  20/40 (68-72 letters) | 1 | 0
  20/32 (73 to 77 letters) | 3 | 0

7. Secondary Outcome: Mean Amblyopic Eye Visual Acuity Letter Scores at 10 Weeks After Stopping Levodopa
Description: as for outcome 5
Time Frame: 10 weeks after stopping levodopa
Measure: Mean (Standard Deviation); unit: letters
Arm/Group | Lower Dose 0.51 mg Levodopa/Carbidopa | Higher Dose 0.76 mg Levodopa/Carbidopa
Number analyzed (Participants) | 16 | 17
letters | 60.6 (11.1) | 53.9 (11.4)

8. Primary Outcome: Mean Change in Amblyopic Eye Visual Acuity Letter Scores at 9 Weeks After Starting Levodopa
Description: as for outcome 3
Time Frame: baseline to 9 weeks
Measure: Mean (Standard Deviation); unit: letters
Arm/Group | Lower Dose 0.51 mg Levodopa/Carbidopa | Higher Dose 0.76 mg Levodopa/Carbidopa
Number analyzed (Participants) | 16 | 17
letters | 3.8 (3.5) | 6.1 (5.6)
Statistical Analysis 1: Comparison: Lower Dose 0.51 mg Levodopa/Carbidopa vs Higher Dose 0.76 mg Levodopa/Carbidopa; Given this was pilot study, no formal sample size estimates were calculated; Test type: Superiority or Other; Mean Difference (Final Values) = -2, 95% CI 2-sided [-6 to 1], Standard Deviation 4.7

9. Primary Outcome: Tolerability of Study Medication-Adverse Event Reporting
Description: Number of adverse events reported throughout entire study.
Time Frame: 24 weeks
Measure: Number; unit: events
Arm/Group | Lower Dose 0.51 mg Levodopa/Carbidopa | Higher Dose 0.76 mg Levodopa/Carbidopa
Number analyzed (Participants) | 16 | 17
events
  Headache | 6 | 6
  Cold/Upper Respiratory Infection/Cough | 3 | 6
  Rash | 1 | 3
  Flu | 2 | 1
  Nausea/Vomiting | 2 | 1
  Fatigue/Sleepiness | 3 | 1
  Dizziness/light-headedness | 3 | 0
  Conjunctivitis | 0 | 2
  Muscle pain | 0 | 2
  Stomach ache | 0 | 2
  Ear ache | 1 | 0
  Fever | 1 | 0
  Loss of appetite | 2 | 0
  Nightmare | 1 | 0
  Knee injury | 1 | 0
  Sinus infection | 1 | 0
  Weight loss | 1 | 0
  Constipation | 1 | 0
  Finger injury | 0 | 1
  Pulled muscle | 0 | 1

10. Secondary Outcome: Distribution of Change in Amblyopic Eye Visual Acuity Scores at 4 Weeks Post Enrollment
Description: as for outcome 3
Time Frame: enrollment to 4 weeks
Measure: Number; unit: participants
Arm/Group | Lower Dose 0.51 mg Levodopa/Carbidopa | Higher Dose 0.76 mg Levodopa/Carbidopa
Number analyzed (Participants) | 16 | 17
participants
  >=15 letters worse | 0 | 0
  10 to 14 letters worse | 0 | 0
  5 to 9 letters worse | 0 | 0
  Within plus or minus 4 letters | 11 | 9
  5 to 9 letters better | 5 | 7
  10 to 14 letters better | 0 | 1
  >=15 letters better | 0 | 0

11. Secondary Outcome: Mean Change in Amblyopic Eye Visual Acuity Letter Scores at 4 Weeks Post Enrollment
Description: as for outcome 3
Time Frame: enrollment to 4 weeks
Measure: Mean (Standard Deviation); unit: letters
Arm/Group | Lower Dose 0.51 mg Levodopa/Carbidopa | Higher Dose 0.76 mg Levodopa/Carbidopa
Number analyzed (Participants) | 16 | 17
letters | 2.9 (2.8) | 3.8 (3.6)

12. Secondary Outcome: Distribution of Change in Amblyopic Eye Visual Acuity Scores at 10 Weeks After Stopping Levodopa
Description: Visual acuity was measured with the electronic early treatment diabetic retinopathy study (E-ETDRS) method and resulted in a letter score that could range from 0 to 97 letters. A difference was calculated as the difference in letters between baseline and outcome with positive difference indicating improvement in acuity.
Time Frame: baseline to 10 weeks after stopping levodopa
Measure: Number; unit: participants
Arm/Group | Lower Dose 0.51 mg Levodopa/Carbidopa | Higher Dose 0.76 mg Levodopa/Carbidopa
Number analyzed (Participants) | 16 | 17
participants
  >=15 letters worse | 0 | 0
  10 to 14 letters worse | 0 | 0
  5 to 9 letters worse | 0 | 1
  Within plus or minus 4 letters | 7 | 8
  5 to 9 letters better | 6 | 7
  10 to 14 letters better | 2 | 1
  >=15 letters better | 0 | 0

13. Secondary Outcome: Mean Change in Amblyopic Eye Visual Acuity Letter Scores at 10 Weeks After Stopping Levodopa
Description: as for outcome 3
Time Frame: baseline to 10 weeks after stopping levodopa
Measure: Mean (Standard Deviation); unit: letters
Arm/Group | Lower Dose 0.51 mg Levodopa/Carbidopa | Higher Dose 0.76 mg Levodopa/Carbidopa
Number analyzed (Participants) | 16 | 17
letters | 4.9 (3.7) | 3.5 (4.7)

ADVERSE EVENTS:
Time Frame: Up to 6 months
Description: Adverse events were systematically collected at each office visit (4wks post-enrollment, 9 wks after starting levodopa, and 10 wks after stopping levodopa) and on each phone call (2wks and 7wks post-enrollment)throughout the study.
Arm/Group | Lower Dose 0.51 mg Levodopa/Carbidopa | Higher Dose 0.76 mg Levodopa/Carbidopa
Serious Adverse Events (participants affected / at risk) | 0/16 | 0/17
Other Adverse Events (participants affected / at risk) | 8/16 | 11/17
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Lower Dose 0.51 mg Levodopa/Carbidopa (N=16) | Higher Dose 0.76 mg Levodopa/Carbidopa (N=17)
Headache (General disorders) | 3 (6) | 3 (6)
Cold/Upper Respiratory Infection/Cough (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 3 (6)
Rash (Skin and subcutaneous tissue disorders) | 1 (1) | 3 (3)
Flu (General disorders) | 2 (2) | 1 (1)
Nausea/Vomiting (Gastrointestinal disorders) | 2 (2) | 1 (1)
Fatique/Sleepiness (General disorders) | 2 (3) | 1 (1)
Dizziness/Light-headedness (General disorders) | 1 (3) | 0 (0)
Conjunctivitis (Eye disorders) | 0 (0) | 1 (2)
Muscle Pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (2)
Stomache Ache (Gastrointestinal disorders) | 0 (0) | 2 (2)
Ear Ache (Ear and labyrinth disorders) | 1 (1) | 0 (0)
Fever (General disorders) | 1 (1) | 0 (0)
Loss of Appetite (General disorders) | 1 (2) | 0 (0)
Nightmare (General disorders) | 1 (1) | 0 (0)
Knee Injury (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Sinus Infection (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Weight Loss (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Constipation (Gastrointestinal disorders) | 1 (1) | 0 (0)
Finger injury (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Pulled Muscle (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)

LIMITATIONS AND CAVEATS:
Without a patching-only control group, no conclusions can be made regarding efficacy, safety, or side effects with this treatment. Placebo controlled trial is needed to see if levodopa can augment occlusion therapy in the treatment of amblyopia.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No